CLINICAL TRIAL: NCT02390011
Title: A Pilot Study of Novel Magnetic Resonance Coil Arrays to Improve the Characterization of Liver Metastases in Patients With Advanced Solid Tumor Malignancies
Brief Title: Pilot Study of Coil Arrays in Patients With Advanced Solid Tumor Malignancies
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 149516
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Neoplams
Keywords: Advanced Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MRI: Day 1
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI

SUMMARY:
This is a single center pilot study testing the use of novel coil arrays with MR liver imaging. In part A of the study, up to 30 healthy volunteers will be scanned, with iterative adjustment of coil array geometry and design to optimize imaging characterstics. In Part B of the study, 40 patients with advanced solid tumors and at least one liver metastasis measuring > 1.5 cm in diameter on standard anatomic scans will undergo MR liver imaging with the newly designed coil array, with the use of gadolinium contrast. Patients with liver tumors will have the option of undergoing a second MR liver scan during the course of subsequent systemic therapy.

ELIGIBILITY:
Inclusion Criteria (Part B only - Patients with advanced solid tumor):

* Advanced solid tumor malignancy and the presence of at least one liver metastasis measuring > 1.5 cm in longest diameter in axial dimension on standard anatomic imaging

Exclusion Criteria (Part B only):

* Contra-indication to gadolinium contrast (e.g. chronic renal disease, prior allergic reaction) for patient studies

Exclusion Criteria (Part A [Healthy Volunteers] and Part B):

* Contra-indication to MRI (e.g. pacemaker, severe claustrophobia, suspected presence of MR-Unsafe surgical implants or shrapnel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Advanced Solid Tumor Malignancies
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2015-05-16 (Actual); Study Completion 2015-05-16 (Actual)

PRIMARY OUTCOMES:
Spatial Resolution | Day 1
  Adjust the coil array to optimize spatial resolution in healthy volunteers
Scan coverage | Day 1
  Adjust the coil array to optimize scan coverage of the liver in healthy volunteers
Mean contrast-to-noise ratio | Day 1
  Detectable using the coil array

SECONDARY OUTCOMES:
Minimum size of detectable metastatic lesion | Day 1
  Detected by MRI scan
Degree signal | Day 1
  Detected by gandolinium contrast in MRI scan within liver metastases
Time-to-peak signal | Day 1
  Detected by gandolinium contrast in MRI scan within liver metastases

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States